CLINICAL TRIAL: NCT05087303
Title: Telemedicine for Pediatric Sickle Cell Patients in Medically Underserved Areas
Brief Title: Telemedicine for Children With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Seethal Jacob, MD, MS, Assistant Professor of Pediatrics, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2101344406; 1K23HL143162-01A1 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-10-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hub and Spoke (Active Comparator)
  Interventions: Other: Types of Telemedicine Delivery Models
- Direct to Consumer (Active Comparator)
  Interventions: Other: Types of Telemedicine Delivery Models

INTERVENTIONS:
Other: Types of Telemedicine Delivery Models — Each arm delivers standard sickle cell care using a different model based on patient location.

SUMMARY:
The purpose of this study is to learn more about how the use of two different types of telemedicine (distance medical care) can address barriers to receiving comprehensive sickle cell care, and whether care can be improved. Aim 1: Adapt two telemedicine models (i.e., hub-and-spoke; direct-to-consumer) for use with children with SCD using caregiver input from our preliminary K12 work. Aim 2: Demonstrate the feasibility of the telemedicine models developed in Aim 1 as the models undergo successive stakeholder refinement during use in actual clinical care. Aim 3: Evaluate the effectiveness of the refined models from Aim 2 in a pre/post study by assessing (a) process of care measures, (b) provider satisfaction, (c) caregiver/patient-centered outcomes, and (d) clinical outcomes and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers must be 18 years or older, who have children between 0 to 21 years old with a diagnosis of Sickle Cell Disease and receive care at the Riley Hospital for Children Comprehensive Sickle Cell Disease clinic.
* Adolescent patients 16 years and older are also able to participate in interviews/surveys.
* The family must be willing to receive their care using the telemedicine model available to them based on the location of their primary residence.
* TeleSCD model participants must live within 1 hour of the pre-identified telemedicine sites, while VirtualSCD model participants must live within the city limits of the pre-identified area.

Exclusion Criteria:

* If a patient receives chronic transfusion therapy, they will not be eligible to participate, as our telemedicine models will not support this.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Measuring adherence to appointment in sickle cell care. | 1 year
  Failed appointments in Electronic Medical Record - no more than one failed appointment during pilot year.
Measuring adherence to lab draws in sickle cell care. | 6 months
  Adherence to lab draws - a minimum of one complete blood count per six months.
Measuring healthcare utilization pre and post telemedicine participation. | 1 year
  Will determine the frequency of 1) vasoocclusive pain episode; 2) acute chest syndrome; 3) Emergency department visits; 4) hospitalizations. This data will be collected through chart abstraction from Electronic Medical Record one year prior to study entry and one year on study.
Measuring collaboration of primary care provider and subspecialty care provider. | 1 year
  Documentation of Primary Care Provider communication of visits in the electronic medical record at least 70% of the time.
Provider Feedback | 1 year
  Telemedicine Acceptance Questionnaire (TAQ) - will be given to all providers participating in telemedicine visits after every telemedicine visit. 0-5 Likert scale
Caregiver feedback | 1 year
  Telemedicine satisfaction survey (TESS) - administered to caregivers following each telemedicine visit. 0-5 Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Seethal Jacob, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States